CLINICAL TRIAL: NCT04106310
Title: The Comparison of Expanded Dialysis With Theranova Dialyzer With Conventional High-flux Hemodialysis
Brief Title: Theranova vs High-flux HD Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Mok Ming Yee, Principal investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1 13th Aug 2019
Record Dates: First submitted 2019-09-10; First posted 2019-09-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The dialyzer used will be covered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theranova (Active Comparator): Patients will be receiving hemodialysis using Theranova dialyzer. The other hemodialysis parameters are kept the same.
  Interventions: Device: Theranova dialyzer
- High-flux (Active Comparator): Patients will be receiving hemodialysis using a high-flux dialyzer. The other hemodialysis parameters are kept the same
  Interventions: Device: High-flux dialyzer

INTERVENTIONS:
Device: High-flux dialyzer — a dialyzer meeting the definition of high-flux
  Arms: High-flux
Device: Theranova dialyzer — a middle cut-off dialyzer
  Arms: Theranova

SUMMARY:
This research proposal of an investigator-initiated clinical study aims to examine the impact of uremic toxin removal afforded by middle cut-off (MCO) dialysis on clinical parameters and surrogate biomarkers pertinent to nutritional, systemic and vascular complications in dialysis patients. The primary research goal is to evaluate the outcomes indicative of nutritional status (as measured by body mass index, body composition monitoring, albumin, clinical assessments such as subjective global assessment, etc.) and parameters relevant to pathophysiological processes in uremia focusing on inflammation and cardiovascular risks. The secondary research aims are to examine dialysis efficacy between MCO dialysis and conventional hemodialysis (CHD). Specifically, dialysis efficacy will be determined by within and between subject differences in baseline versus short term (6 months) and long term (12 months) effects of MCO dialysis and CHD in:

1. Removal of small molecules (e.g. urea), middle molecules (Beta-2 microglobulin, Phosphate and Creatinine) and protein bound solutes
2. Markers of inflammation, ossification and fibrosis
3. Uremia associated epigenetic modification The investigators hypothesize superiority of nutritional parameters in patients undergoing MCO dialysis compared with patients on CHD. The investigators plan to randomize 60 patients to either MCO dialysis or CHD at two hemodialysis units in Hong Kong.

DETAILED DESCRIPTION:
Accumulation of uremic toxins is associated morbidity and mortality in patients with end-stage renal disease, but the pathogenic mechanisms how they lead to various clinical complications remain elusive. Conventional hemodialysis is effective in removing small molecular solutes (in the range of 50-15,000 Da), but the removal of protein-bound and middle to larger molecular toxins (up to 50,000 Da) remains unsatisfactory even with augmented hemodialysis frequency or duration. The notion that dialysis adequacy is no longer a simple quantitative measure of small molecular removal has led to the clinical application of intensive hemodialysis and the search for novel strategies to reduce uremic toxin burden.

Recently, a new class of membrane with molecular weight cut off (MWCO) close to the molecular weight of albumin was introduced. The focus of this new therapy, known as expanded dialysis using the medium cut off (MCO) dialysis membrane, is to provide the potential for more efficient removal of middle molecules and protein bound uremic toxins without excessive loss of albumin. To date, MCO dialysis has been associated with a reduction in transcription of pro-inflammatory cytokines (i.e. interleukin 6 and tumor necrosis factor-α) and middle molecules especially free lambda light chains.

Protein-energy wasting and cardiovascular diseases are prevalent in chronic kidney disease and is related to inflammation and increased mortality. Despite growing data on the clearance of individual uremic toxins and biochemical parameters, the impact of MCO dialysis on clinical outcomes and mechanistic parameters related to nutrition and inflammation remains to be investigated.

The objective of the study is to compare MCO dialysis with conventional high-flux HD, on nutritional parameters, inflammation and cardiovascular biomarkers and related clinical outcomes.

Since twice-weekly HD is commonly practiced in Hong Kong, this study provides a distinct opportunity to investigate whether MCO dialysis might be particularly advantageous in patients receiving a relatively lower dialysis dose through the removal of a broader spectrum of uremic toxins.

The investigators hypothesize that MCO dialysis with Theranova Dialyzer (HDx) improves parameters related to nutrition and inflammation compared with high-flux HD.

This will be a prospective single-blinded, randomized, controlled trial with stable HD patients randomized at 1:1 ratio to either one of the following - A. to continue with HD using the same high-flux dialyzer as in the previous 6 weeks (high-flux HD arm) B. change to HDx using Theranova Dialyzer (MCO dialysis arm)

ELIGIBILITY:
Inclusion Criteria:

* adult patients age greater than 18 years old
* end-stage renal failure on two- or three-times per week high-flux HD for more than 90 days
* mean spKt/Vurea >1.2 per session (for 3 dialysis sessions per week) or spKt/Vurea >1.8 per session (for 2 dialysis sessions per week)

Exclusion Criteria:

* active malignancy
* unable to give informed consent or complete questionnaires
* unstable clinical condition defined as significant clinical event requiring hospitalization in the past 90 days
* unreliable vascular access
* unable to achieve HD blood flow >150ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
lean tissue index | 12 months
  measured by Body Composition Monitor
Body Mass Index | 12 months
  measured by weight (in kilograms) divided by the square of heights (in meters)

SECONDARY OUTCOMES:
asymmetrical dimethylarginine | 12 months
  endogenous inhibitor of nitric oxide synthase, one of the cardiovascular biomarkers
fibroblast growth factor 23 | 12 months
  biomarker for bone turnover
Klotho | 12 months
  biomarker for atherosclerosis and bone turnover
Kt/V urea | 12 months
  measurement of clearance of urea by hemodialysis therapy, a marker for adequacy of dialysis
beta-2 microglobulin | 12 months
  middle size uremic toxin
Pentraxin-3 | 12 months
  middle to large molecular size uremic toxin
soluble endothelial protein C receptor | 12 months
  a marker for endothelial dysfunction
soluble thrombomodulin | 12 months
  a marker for endothelial dysfunction
hemoglobulin | 12 months
  indication of anemia
high-sensitive C reactive protein | 12 months
  marker for inflammation
interleukin 6 | 12 months
  marker for inflammation
tumor necrosis factor alpha | 12 months
  marker for inflammation
albumin | 12 months
  marker for nutritional status
Leptin | 12 months
  marker for nutritional status and appetite
adiponectin | 12 months
  nutritional marker
phosphate | 12 months
  small size uremic waste produce
low-density lipoprotein | 12 months
  reflects lipid control
high-density lipoprotein | 12 months
  reflects lipid control
triglyceride | 12 months
  reflects lipid control
Malnutrition-Inflammation Score | 12 months
  a measurement scale reflecting nutritional status
Subjective Global Assesment questionnaire | 12 months
  a measurement scale reflecting nutritional status
fat tissue index | 12 months
  nutritional marker measured by Body Composition Monitor
admission rate due to cardiovascular events | 12 months
  number of admisisons due to cardiovascular events during the follow-up period
admission rate due to infection | 12 months
  number of admissions due to infection during the follow-up period
mortality rate | 12 months
  number of deaths during the follow-up period
5-D itch scale | 12 months
  Symptomatology scale to measure itchiness
Numeric rating scale for itchiness | 12 months
  Symptomatology scale to measure itchiness
The Functional Assessment of Anorexia/Cachexia Therapy (FAACT) score | 12 months
  measurement scale for appetite
Visual analogue scale for appetite | 12 months
  measurement scale for appetite
Postdialysis recovery time | 12 months
  number of time required to feel well after receiving a hemodialysis session
Self-reported sleep quality | 12 months
  scale to rate the quality of sleep
Hong Kong Montreal Cognitive Assessment | 12 months
  measurement of cognitive function
KDQOLSFTMv1.3 questionnaire | 12 months
  quality of life assessment
DNA methylation analysis of TRPV1 gene | 12 months
  epigenetics modification
DNA methylation analysis of LY96 gene | 12 months
  epigenetics modificaiton
DNA methylation analysis of IFNGR1 gene | 12 months
  epigenetics modifications

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Ming Yee Mok, MBBS, MRCP, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Division of Nephrology, Department of Medicine, Queen Mary Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mok MMY, Yung S, Kwan LPY, Yip TPS, Lui SL, Chan TM. Expanded Hemodialysis with Theranova Compared with Conventional High-Flux Hemodialysis: Prospective Randomized 12-Month Study. Kidney360. 2025 Mar 18;6(7):1143-1157. doi: 10.34067/KID.0000000769. PMID 40100276